CLINICAL TRIAL: NCT02695511
Title: CALERIE Phase II Ancillary 2: Metabolic Adaptation After Two Years of Caloric Restriction in Non Obese Humans
Brief Title: CALERIE Phase II Ancillary: Metabolic
Acronym: CALERIE-II
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pennington Biomedical Research Center (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Eric Ravussin, Principal Investigator, Pennington Biomedical Research Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PBRC 26039-A; R01AG029914 (NIH)
Record Dates: First submitted 2016-01-13; First posted 2016-03-01 (Estimated); Last update posted 2016-03-01 (Estimated); Status verified 2016-02

CONDITIONS: Aging
MeSH Terms: interventions — Caloric Restriction

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 25% CR (Experimental): 25% caloric restriction
  Interventions: Other: Caloric restriction
- CO (control) (No Intervention): healthy lifestyle recommendation

INTERVENTIONS:
Other: Caloric restriction — 25% caloric restriction below baseline energy requirement
  Arms: 25% CR

SUMMARY:
The primary aim of this NIA sponsored ancillary study of phase 2 CALERIE is to measure whether metabolic adaptation lasts up to 2 years in response to a 25% calorie restriction in normal-weight and slightly overweight individuals. Energy metabolism (24-hour sedentary and sleeping) will be measured in a respiratory chamber. Other measures include the activities of the sympathetic nervous and thyroid axes, oxidative stress in lipids, protein and DNA, organ size by MRI and echocardiography, and posture allocation (time spent engaging in different activities and the energy expended during these activities), and activity temperament (the innate predilection for movement). This set of studies will allow assessment of whether the previously observed metabolic adaptation in response to 25% caloric restriction is long lasting (up to two years), associated with reduced thyroid and sympathetic activities and reduced oxidative damage. The studies of organ sizes (liver, spleen, kidney, heart, adipose and muscle) by MRI and echo (heart) is essential to determine whether the metabolic adaptation is related to decreased organ sizes or improved organ energy metabolism efficiency. The above described measures will be performed at baseline and after 1 and 2 years of a 25% caloric restriction in 50 non-obese humans and in 25 sex-, BMI- and age- matched subjects who will not engage in caloric restriction.

DETAILED DESCRIPTION:
Hypothesis 1: The decrease in energy expenditure (sedentary and sleeping) will be larger than that expected on the basis of loss of fat-free mass and fat mass even after weight stabilization. Aim 1: Determine the metabolic adaptation after 1 and 2 years of a 25% CR

Hypothesis 2: The metabolic adaptation (what is not accounted by a decrease in FM and FFM) is not entirely accounted by reduced organ/tissue size (liver, spleen, kidney, heart and brain) but is accompanied by reduced activities of the sympathetic and thyroid systems. Aim 2: Assess the contribution of organ sizes and activities of the thyroid and sympathetic systems to the metabolic adaptation. Results will be compared to in vivo and in vitro oxidative phosphorylation (Smith, PI).

Hypothesis 3: A decrease in markers of oxidative stress to lipid (urinary isoprostanes) DNA (strand breaks) in blood and protein (carbonylation and thiol oxidation) in blood and skeletal muscle tissue after 1 and 2 years of CR will be observed. Aim 3: Determine the changes in oxidative stress after 1 and 2 years of 25% CR by measuring urinary isoprostanes, serum carbonyls, DNA damage in nucleated blood cells and protein oxidation (carbonyls and oxidation of cysteine residues) in skeletal muscle.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and women
* > 22 BMI < 28 kg/m2
* > 25 age < 46

Exclusion Criteria:

* History or clinical manifestation of cardiovascular disease or an elevated blood pressure (greater than 140/90 mm Hg)
* Abnormal resting ECG
* History or clinical manifestation of diabetes, cholelithiasis or any other significant metabolic, hematologic, pulmonary, cardiovascular, gastrointestinal, neurologic, immune, hepatic, renal, urologic disorders, eating disorders or cancer
* History of stomach or intestinal surgery (except appendectomy) or major abdominal, thoracic or non-peripheral vascular surgery within one year prior to the randomization date
* Any disease or condition that seriously affects body weight and/or body composition
* Potassium level above the upper limit of normal at the screening visit confirmed by a test repeated within two weeks
* Hemoglobin, hematocrit, RBC, or iron level below the lower limit of normal at the screening visit confirmed by a test repeated within two weeks
* Evidence of active liver disease or ALT levels above 1.5 times the upper limit of normal
* Any history of pharmacologic treatment for a psychiatric disorder within one year prior to the randomization date or a history of more than one episode of a pharmacologic treatment for a psychiatric disorder within lifetime
* History of drug or alcohol abuse (up to 14 drinks a week are allowed) within the past two years
* Individuals who present with a BDI score of =15 at screening or baseline
* Short-term (less than a month) treatment with steroids within six months prior to the randomization date
* Treatment with steroids for more than a month within five years prior to the randomization date
* Regular use of other medications, except oral contraceptives
* Individuals who participated in the CALERIE Phase 1 studies
* A volunteer must be either be a never-smoker of tobacco products or an ex-smoker who quit completely at least 12 months prior to the screening visit
* Individuals who have magnetic metallic objects in their body
* Individuals who donated blood within 30 days prior to the randomization date
* Concurrent participation in any other interventional study
* Pregnant or breast-feeding women
* Individuals who were engaged in a regular program of physical fitness involving some kind of heavy physical activity (e.g., jogging, running or riding fast on a bicycle for 30 minutes or more) five or more times per week over the past year
* Unwilling to be assigned at random to the CR or control intervention
* Unwilling or unable to adhere to the rigors of the CR intervention over the entire two-year intervention
* Individuals who unable or unwilling to discontinue dietary supplements or adhere to the alcohol consumption restrictions during the study
* Unwilling or unable to adhere to the rigors of the data collection and clinical evaluation schedule

Ages: 25 Years to 46 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 75 (Actual)
Dates: Start 2007-05; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Change in 24-h Sedentary Energy Expenditure from Baseline | Baseline, 1 and 2 years
  Measured via Respiratory Chamber
Change in 24-h Sleeping Energy Expenditure from Baseline | Baseline, 1 and 2 years
  Measured via Respiratory Chamber

SECONDARY OUTCOMES:
Change in Oxidative Stress from Baseline | Baseline, 1 and 2 years
Change in Organ/Tissue Size from Baseline | Baseline, 1 and 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Eric Ravussin, PhD, Principal Investigator — Pennington Biomedical Research Center
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Shen W, Chen J, Zhou J, Martin CK, Ravussin E, Redman LM. Effect of 2-year caloric restriction on organ and tissue size in nonobese 21- to 50-year-old adults in a randomized clinical trial: the CALERIE study. Am J Clin Nutr. 2021 Oct 4;114(4):1295-1303. doi: 10.1093/ajcn/nqab205. PMID 34159359
- [Derived] Broskey NT, Marlatt KL, Most J, Erickson ML, Irving BA, Redman LM. The Panacea of Human Aging: Calorie Restriction Versus Exercise. Exerc Sport Sci Rev. 2019 Jul;47(3):169-175. doi: 10.1249/JES.0000000000000193. PMID 30998529
- [Derived] Redman LM, Smith SR, Burton JH, Martin CK, Il'yasova D, Ravussin E. Metabolic Slowing and Reduced Oxidative Damage with Sustained Caloric Restriction Support the Rate of Living and Oxidative Damage Theories of Aging. Cell Metab. 2018 Apr 3;27(4):805-815.e4. doi: 10.1016/j.cmet.2018.02.019. Epub 2018 Mar 22. PMID 29576535
- [Derived] Sparks LM, Redman LM, Conley KE, Harper ME, Yi F, Hodges A, Eroshkin A, Costford SR, Gabriel ME, Shook C, Cornnell HH, Ravussin E, Smith SR. Effects of 12 Months of Caloric Restriction on Muscle Mitochondrial Function in Healthy Individuals. J Clin Endocrinol Metab. 2017 Jan 1;102(1):111-121. doi: 10.1210/jc.2016-3211. PMID 27778643